CLINICAL TRIAL: NCT01807936
Title: Esophagectomy: Three-field Lymphadenectomy Versus. Two-field Lymphadenectomy for Thoracic Middle and Lower Esophageal Cancer
Brief Title: Esophagectomy:Three-field Versus Two-field Lymphadenectomy (ECTOP-2002)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Fudan University cancer hospital, Fudan University cancer hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2VS3E
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Esophageal Neoplasms
Keywords: Esophageal Neoplasms; lymphadenectomy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Three-field lymphadenectomy (Experimental): Cervical-thoracic-upper abdominal three-field lymphadenectomy
  Interventions: Procedure: Lymphadenectomy
- Two -field lymphadenectomy (No Intervention): Thoracic-upper abdominal two -field lymphadenectomy

INTERVENTIONS:
Procedure: Lymphadenectomy
  Arms: Three-field lymphadenectomy

SUMMARY:
This is a clinical trial from Eastern Cooperative Thoracic Oncology Project (ECTOP), numbered as ECTOP-2002. Esophageal carcinoma is an aggressive disease with a poor prognosis. Surgical resection with radical lymphadenectomy remains the basic method of management of this malignancy. Lymph node metastasis is one of the most important factors in predicting the prognosis of patients with esophageal carcinoma, but the extent of lymph node dissection is still in debate, and there is no statistical evidence based on large scale prospective randomized trials with regard to the issue that which is the optimal extent of lymphadenectomy for esophageal cancer. The purpose of this study is to test two different extents of lymphadenectomy (Cervical-thoracic-upper abdominal three-field lymphadenectomy and Thoracic-upper abdominal two -field lymphadenectomy) in middle or lower third intrathoracic esophageal cancer. This research is being done to see whether one extent of lymphadenectomy is superior than the other with better long-term outcome and acceptable postoperative short-term outcome or not.

DETAILED DESCRIPTION:
Background :

Esophageal carcinoma is an aggressive disease with a poor prognosis. Surgical resection with radical lymphadenectomy remains the basic method of management of this malignancy. The international Society for Diseases of the Esophagus has classified the extent of lymphadenectomy as standard, extended, total, and three-field lymphadenectomy. However, lymph node metastases can be present as regional metastasis, skip metastasis and distant metastasis, the optimal extent of lymphadenectomy remains controversial by now. Three-filed lymphadenectomy was criticized for higher surgical risks, but have the merits of removing all potential positive nodes and reducing the local recurrence. The purpose of this study is to conduct a large scale prospective randomized Phase Ⅲ clinical trial to test that based on the long-term outcomes(overall survival and disease free survival )and postoperative short-term outcomes(mortality, morbidity),whether one extent of lymphadenectomy is superior than the other approach or not.

Objectives:

1. To compare overall survival after three-field lymphadenectomy and two-field lymphadenectomy
2. To compare locoregional recurrence, disease free survival after three-field lymphadenectomy and two-field lymphadenectomy
3. To compare postoperative morbidity and mortality in the two groups

Design: Prospective randomized controlled Setting: Fudan University Cancer Center, Shanghai, China. Patients and methods : All patients with biopsy proven carcinoma of the middle or lower third of the esophagus presenting to our hospital will be considered for the study.

Staging investigations will be standard and will include

1. Computed Tomography (CT) scans in all patients
2. Esophagogastroscopy
3. Barium swallow
4. Endoscopic Ultrasonography (EUS) wherever possible
5. PET-CT scan wherever possible

Randomization:

Randomization, by the sealed envelope method, took place on the morning of planed surgery day.

All surgeries will be performed under general anesthesia with epidural analgesia. The surgery will be either performed by or under the direct supervision of consultant thoracic surgeons with experience in esophageal surgery. Operative time, blood loss, blood product replacement and all intraoperative details will be recorded in the proforma. Patients will be shifted postoperatively to the intensive care unit (ICU) for observation and subsequently to the recovery or high dependency ward once stabilized. Postoperative details including period of postoperative ventilation, hemorrhage, pulmonary and cardiac complications, arrhythmias, thoracic duct leak, anastomotic leak, wound infection and recurrent laryngeal nerve paresis or palsy will be recorded. Postoperative mortality will be defined as 30-day mortality plus death before discharge after surgery. The total duration of ICU stay and hospital stay will also be recorded.

Follow up:

Patients will be followed up three monthly for the first two years and six monthly for the third to fifth years and annually thereafter. A detailed history and clinical examination and CT scan, barium swallow and ultrasound will be done routinely on every follow up.

Data management: All collected data will be entered into a statistical software package for subsequent analysis

Main research variables:

Primary end point: Overall survival

Secondary endpoints:

1. Disease free survival in the two arms
2. Locoregional recurrence
3. Postoperative morbidity and mortality

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven squamous cell esophageal cancer
* Patients with cT1-T3/N0-N1 mid or distal third (inferior to carina and 3cm superior to cardia ) operable esophageal lesion. Staging investigations including esophagogastroscopy, chest and abdominal CT scan, barium swallow and selective endoscopic ultrasonography showing no evidence of invading adjacent structure such as spine, bronchus, pericardium , descending aorta and without enlargement cervical and celiac nodes (diameter of short axis greater than 1.5cm) measured at CT scans.
* Karnofsky performance status greater than or equal to 80%
* Pulmonary and cardiac function must be acceptable for surgery according to institutional standards.
* Acceptable hepatic, renal and bone marrow function

Exclusion Criteria:

* Patients with low performance status(Karnofsky score <80%)
* Past history of malignancy
* Stage investigations indicating unresectable advanced disease(T4 or M1a,M1b)
* Patients with any other serious underlying medical condition that would impair the ability of the patient to receive or comply with protocol treatment
* Patients medically unfit for surgical resection
* Patients with pulmonary reserve inadequate to undergo thoracotomy and extensive mediastinal lymphadenectomy.
* Patients with a significant history of unstable cardiovascular disease that in the opinion of the treating physician should preclude the patient from protocol treatment.
* Uncontrolled diabetes mellitus or uncontrolled infection, including HIV or interstitial pneumonia or interstitial fibrosis.
* Significant psychiatric illness that would interfere with patient compliance
* Patients with severe hepatic cirrhosis or with serious renal disease unacceptable for surgery
* Patients considered of salvage surgery after definitive chemoradiotherapy
* Patients after neoadjuvant chemoradiotherapy
* Patients above the age of 75 years
* Patients unreliable for follow up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-03-20 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years.
  Participants will be seen at regular interval of 3 months the first year and every 6 months until death or the 3rd year.

SECONDARY OUTCOMES:
Disease free survival | 3 years
  Participants will be seen at regular interval of 3 months the first year and every 6 months until recurrence or the 3rd year.

OTHER OUTCOMES:
postoperative morbidity and mortality | an average of 2 weeks
  Participants will be followed for the duration of hospital stay. An average of hospital stay was 2 weeks.
locoregional recurrence and recurrence pattern | 3 years
  Participants will be seen at regular interval of 3 months the first year and every 6 months until recurrence or the 3rd year.

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li B, Hu H, Zhang Y, Zhang J, Miao L, Ma L, Luo X, Zhang Y, Ye T, Li H, Li Y, Shen L, Zhao K, Fan M, Zhu Z, Wang J, Xu J, Deng Y, Lu Q, Li H, Zhang Y, Pan Y, Liu S, Hu H, Shao L, Sun Y, Xiang J, Chen H. Three-field versus two-field lymphadenectomy in transthoracic oesophagectomy for oesophageal squamous cell carcinoma: short-term outcomes of a randomized clinical trial. Br J Surg. 2020 May;107(6):647-654. doi: 10.1002/bjs.11497. Epub 2020 Feb 28. PMID 32108326